CLINICAL TRIAL: NCT06210022
Title: Cognitive Impairment in Drug-resistant and Drug-responsive Focal Cryptogenic Epilepsy: a Longitudinal Observational Study
Brief Title: Cognitive Impairment in Drug-resistant and Drug-responsive Focal Cryptogenic Epilepsy
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Prof. Massimo Filippi, Professor Massimo Filippi, IRCCS San Raffaele
Other Study IDs: FCECOG
Record Dates: First submitted 2023-12-21; First posted 2024-01-18 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Epilepsy; Focal Epilepsy
Keywords: epilepsy; focal cryptogenic epilepsy; drug resistant epilepsy
MeSH Terms: conditions — Epilepsy; Epilepsies, Partial; Drug Resistant Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 130: Patients with diagnosis of DRE and DSE will be recruited among patients who are regularly followed at our Epilepsy Outpatients Service (OSR). The diagnosis of DRE and DSE focal cryptogenic epilepsy will be based on the most recent sets of criteria of different types of epilepsy. A small group of NDE patients will be also enrolled
  A population of 30 focal cryptogenic epilepsy patients diagnosed with DRE (drug resistant epilepsy) A population of 90 focal cryptogenic epilepsy patients diagnosed with DRE (drug sensitive epilepsy) 10 patients newly diagnosed for focal cryptogenic epilepsy (NDE) will be recruited too.
  Interventions: Diagnostic Test: Neuropsychological Assessment

INTERVENTIONS:
Diagnostic Test: Neuropsychological Assessment — Cognitive evaluation and clinical monitoring of seizure frequency

SUMMARY:
This is a national monocentric (San Raffaele Hospital - OSR, Via Olgettina, 60, 20132 Milan, Italy) observational low-risk-intervention study, prospective and multiparametric (clinical, EEG, neuropsychological evaluations) study.

Patients with a diagnosis of DRE and DSE will be screened to evaluate their eligibility. They will undergo clinical and cognitive assessments in addition to 32channel EEG at baseline (T0). DRE patients will also undergo clinical and cognitive assessments, and 32-channel EEG at 6 months (T1), and 12 months (T2). Patients newly diagnosed with focal cryptogenic epilepsy (NDE) will undergo clinical and cognitive assessments, and 32-channel EEG at baseline (T0), at 6 months (T1), and 12 months (T2).

High-definition EEG will be performed to investigate patterns of cortical sources and functional connectivity alteration specific to DRE and DSE and to explore their prognostic value. Longitudinal EEGs will be acquired to explore the evolution of EEG patterns.

Cognitive evaluation will be performed by an experienced neuropsychologist. At baseline, DRE, DSE, and NDE patients will undergo a screening and a comprehensive cognitive battery in order to define performance differences among groups. The DRE and NDE group only will perform the same neuropsychological assessment at month 6 and 12 for monitoring the potential progression of cognitive and/or behavioural disturbances in these patients.

DETAILED DESCRIPTION:
At the study entry (T0) DSE, DRE, and NDE will undergo cognitive evaluations (investigating the main cognitive domains), neurological examinations, and 32channel EEG. DRE and NDE patients will undergo the same clinical, cognitive and 32-channel EEG evaluations at T1 (6 months) and T2 (12 months). DSE patients will be tested only at baseline and they will not undergo longitudinal evaluations.

ASM therapy and seizure frequency will be recorded for DRE and NDE patients in a dedicated database at T0, T1 and T2 High-density EEGs, with a duration of 20 minutes, will be acquired in resting awake conditions on a computer-based system (Micromed System PLUS, Micromed S.p.A., Mogliano Veneto, Italy) from 32 surface electrodes, placed on an EEG cap according to the international 10/20 system, with linked-ear or mesial prefrontal reference. Vigilance will be continuously monitored in order to avoid drowsiness. The quality of sleep during the night previous to the exam will be investigated by the recording technician. Standard clinical procedures will be implemented in the acquisition protocol.

Cognitive evaluations will be performed by an experienced neuropsychologist. The following domains will be assessed: global cognition, memory, language, attention, executive functions, visuospatial abilities, mood and behavior. Moreover, for the assessment of quality of life, the 12-item Short Form Survey (SF-12) will be administered to DSE patients at baseline, and to NDE patients and DRE at baseline and at the follow-up.

Clinical and cognitive data will be exported and analyzed through SPSS and/or R software afterwards. All demographic, personal and clinical information will be codified.

EEG will be stored in a digital archive and on CDs, and then uploaded on dedicated PCs and Linux stations in order to perform the analyses

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for all study subjects:

  * monolingual native Italian speakers;
  * age between 18-60 years;
  * normal or corrected-to-normal visual acuity;
  * oral and written informed consent to study participation.
  * if assuming psychotropic drugs (i.e., benzodiazepines, antipsychotics, antidepressants), they should be at stable dosage for more than 4 weeks.
* Inclusion criteria for DRE patients:

  * diagnosis of focal cryptogenic epilepsy;
  * previous failure of at least 2 anti-seizure medication (ASM at adequate dose;
  * at least 3 seizures in the last 2 months; • available brain MRI (<5 years).
* Inclusion criteria for DSE patients:

  * diagnosis of focal cryptogenic epilepsy;
  * seizure control obtained after not more than 2 ASM;
  * seizure freedom for at least 6 months;
  * available brain MRI (<5 years).
* Inclusion criteria for NDE patients:

  * new diagnosis of focal cryptogenic epilepsy (<3 months)
  * not more than 1 ASM tested
  * available brain MRI (<3 months)

Exclusion Criteria:

* Age> 60 years;
* Documented developmental delay;
* Evidence of focal abnormalities at neuroimaging (except of hippocampal sclerosis);
* Neurological degenerative conditions;
* history of other systemic (including systemic neoplasms in the last 3 years and abnormal hepatorenal functions), neurologic, psychiatric diseases, head injury, cardiovascular events, and cerebrovascular alterations;
* alcohol and/or psychotropic drugs abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with diagnosis of DRE and DSE will be recruited among patients who are regularly followed at our Epilepsy Outpatients Service (OSR). The diagnosis of DRE and DSE focal cryptogenic epilepsy will be based on the most recent sets of criteria of different types of epilepsy.
  A small group of NDE patients will be also enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the prevalence of cognitive impairment in a population of focal cryptogenic epilepsy patients, comparing subjects diagnosed with DRE (drug resistant epilepsy) and subjects diagnosed with DSE (drug sensitive epilepsy); | 2024-2027
  At baseline, DRE and DSE patients will undergo a screening and comprehensive cognitive battery. We will adopt the following scales: EpiTrack screening battery; Rey Auditory Verbal Learning Test and with the Rey's figure recall; Token Test; Paced Auditory Serial Addition Test; Modified Card Sorting Test; Cognitive Estimation Task; Rey's figure copy, Beck Depression Inventory, Dimensional Apathy Scale, 12-item Short Form Survey. The suspect of cognitive impairment (CI) will be defined with EpiTrack screening battery (score < 32 points indicates CI). This will be confirmed by the comprehensive battery (Level II): Impairment should be present on at least 2 tests. For each test, impairment will be demonstrated with performances below appropriate normative values. Since the classification for CI is not yet defined for epilepsy we will adopt the classification for Parkinson's disease which, as patients with epilepsy, mainly have disturbances in executive, attentive and memory functioning.
To monitor the evolution of cognitive performance in DRE patients over a period of one year; | 2024-2027
  we evaluate the cognitive state of the patients with the measures and scales listed in "Outcome 1" at 12 months and compare the results to the baseline results.
To evaluate whether seizure frequency constitute the main determinant of cognitive impairment; | 2024-2027
  We evaluate if patients who reduced the seizure frequence over a period of 12 months showed an improvement in the cognitive assesment, comparing baseline assesment and the follow up assesment at 12 months.
To explore EEG-markers of DRE and DSE | 2024-2027
  High-density EEGs, with a duration of 20 minutes, will be acquired in resting awake conditions on a computer-based system (Micromed System PLUS, Micromed S.p.A., Mogliano Veneto, Italy) from 32 surface electrodes, placed on an EEG cap according to the international 10/20 system, with linked-ear or mesial prefrontal reference. Vigilance will be continuously monitored in order to avoid drowsiness.
  EEG will be performed to investigate patterns of cortical sources and functional connectivity alteration in the two different groups od DRE and DSE.
To evaluate the entity of cognitive impairment in a population of focal cryptogenic epilepsy patients, comparing subjects diagnosed with DRE (drug resistant epilepsy) and subjects diagnosed with DSE (drug sensitive epilepsy); | 2024-2027
  To evaluate the entity of cognitive impairment in DSE with the measures and methods specified in "Outcome 1".
To evaluate whether ASM therapy constitute the main determinant of cognitive impairment; | 2024-2027
  We evaluate if patients who reduced the number of ASMs medications over a period of 12 months showed an improvement in the cognitive assesment, comparing baseline assesment and the follow up assesment at 12 months.
To explore a possible relationship between EEG-markers of DRE and DSE and cognitive impairment | 2024-2027
  To explore a possible relationship between EEG-markers of DRE and DSE found as specified in "Outcome 4" and cognitive impairment (evaluated as specified in "Outcome 1").

SECONDARY OUTCOMES:
To evaluate longitudinal evolution of cognitive performances in patients newly diagnosed with focal cryptogenic epilepsy (NDE) | 2024-2027
  At baseline, NDE patients will undergo a screening and a comprehensive cognitive battery in order to define performance differences among groups. The NDE patients groups only will perform the same neuropsychological assessment at month 6 and 12 for monitoring the potential progression of cognitive and/or behavioral disturbances in these patients.
  We will use the same neuropsychological scales listed in "Outcome 1".
To evaluate longitudinal evolution of drug responsiveness in patients newly diagnosed with focal cryptogenic epilepsy (NDE) | 2024-2027
  We evaluate if over a period of 6 and 12 months the patients of NDE groups have showed drug responsiveness, assessed as "reduction of number of seizure per month", compared to the baseline data.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele, Milan, Italy